CLINICAL TRIAL: NCT02522065
Title: Motor Response to Dopaminergic Therapy in a Population of de Novo Parkinson's Disease Cases Quantified Via Typing Analyses - -neuroQWERTY
Brief Title: neuroQWERTY: a Transparent Patient-centered Outcome Method to Quantify Parkinsonian Motor Signs for Drug Trials
Acronym: neuroQWERTY
Status: Completed | Type: Observational
Sponsor: Fundación de investigación HM (Other)
Collaborators: Massachusetts Institute of Technology (Other); Hospital Universitario 12 de Octubre (Other); Hospital San Carlos, Madrid (Other); Hospital Universitario Ramon y Cajal (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Fundación Alcorcón (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: 15.05.796-GHM
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: Hypokinesia; Patient Outcome Assessment
MeSH Terms: conditions — Parkinson Disease; Hypokinesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls: A sample of 30 healthy volunteers will be recruited to compare the typing signal with that of the cases.
- Early Parkinson's disease cases: A sample of 30 early PD cases (i.e. less than five years of disease and no axial signs or fluctuations) that are going to be prescribed de novo dopaminergic therapy will be recruited.

SUMMARY:
The motor impairment produced by Parkinson's disease (PD) is a significant and debilitating part of the condition. Current methods to evaluate this impairment rely on subjective examinations. The investigators seek to develop an objective assessment of motor deficits by monitoring the participants natural interactions with a keyboard (on a computer or smart device). This approach provides a window to how the brain behaves during typical daily use of these devices, i.e. writing a report, sending an email or any other task performed on a digital device and thus has the potential to be used easily and regularly. (Importantly, the data gathered are non-sensitive and based only on timing information).

PD participants will be recruited during outpatient visits to PD clinics throughout the Madrid metropolitan region. General entry criteria will be those patients who are scheduled to begin dopaminergic therapy, and own a home computer or laptop. The study will not impact on participants' standard clinical management other than by asking the participants to type for 15 minutes at each of the clinic visits, and installing the investigators proprietary software on their home computer. This software will collect keystroke data alone. (None of the actual information about what is being typed will be collected.) The keystroke data collected will be analyzed and compared with standard clinical metrics of therapeutic response, as well as the in-clinic typing data.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 18 years and 70 years (older subjects will be deemed eligible on an individual basis after review by the study team).
2. Parkinson's disease (PD) diagnosis according to the United Kingdom Brain Bank Criteria.
3. PD patients without cognitive or psychiatric disturbances, as measured by the baseline assessment.
4. Prescription of symptomatic therapy with L-Dopa or dopamine agonists based on functional impairment attributed to PD. This will be based on the participant's physician criteria based on:

   * Involvement of the dominant hand and/or upper limbs.
   * Employed patients which the disease impairs their ability to work.
5. Daily computer use > 30 minutes

Exclusion Criteria:

1. Mild cognitive impairment or dementia.
2. Psychiatric symptoms
3. Expected or current use of sedative medication (benzodiazepines, opiates, antihistaminergic drugs).
4. Neuroleptic use.
5. History of parkinsonism for the controls.
6. Severe osteo-articular problems with upper limb functional limitation (amputations, severe osteo-arthritis).
7. Alcohol risk use (>40 gr/day or 4 standard drinks for male / >24gr/day or 2 standard drinks for female).
8. Narcolepsy or other sleep disorder producing hypersomnia (obstructive apnea, acute confusional states).
9. Any other life- threatening condition (advanced cancer, severe hepatic or renal insufficiencies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of early Parkinson's disease participants who are going to be prescribed dopaminergic agents and a group of healthy volunteers will be recruited at the different collaborating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a motor response to medication > 4 UPDRS-III points detected by the developed algorithm (sensitivity to a motor change). | 24-weeks
  A diagnostic table will be computed with all the study subjects. Those subjects with a clinical relevant response to medication (> 4 points in UPDRS - III) will be considered as true positives. Then, the accuracy of the typing test to detect them will be evaluated. For this purpose, the sensitivity, specificity, predictive values and ROC curve of a classification algorithm based on our nQ index will be computed. This will allow us assessing the validity of the test to identify a motor change. detected by the developed algorithm (sensitivity to a motor change).

SECONDARY OUTCOMES:
Agreement between nQ and UPDRS motor subscale | 4,8,16,24-weeks
  Correlation (Spearman Rho) analyses between the indices and UPDRS
Comparison between nQ and the different motor tests (Purdue Pegboard test score & Alternating Finger Tapping) | 4,8,16,24-weeks
  Correlation (Spearman Rho) between the indices and motor test scores
Effect of dopaminergic medication measured by nQ | 4,8,16,24-weeks
  Correlation (Spearman Rho) between the indices and drug titration measured in L-Dopa equivalent milligrams
Comparison between nQ and the CISI-PD, PDQ-39 and NMSS scales | 4,8,16,24-weeks
  Correlation (Spearman Rho) between the indices and the CISI-PD, PDQ-39 and NMSS scales.
Stability of the nQ index in a less controlled environment ("home-setting"). | Week 1
  Bland-Altman analyses to evaluate the stability of the indices in different days where the medication was not changed and therefore a change should not be expected

CONTACTS AND LOCATIONS:
Overall Officials: Jose Obeso, MD, PhD, Principal Investigator — Director at Centro Integral de Neurociencias A.C.
Locations (6):
- Spain (6):
  - Fundacion Hospital Alcorcón, Alcorcón, Madrid
  - Hospital Universitario HM Puerta del Sur - Centro Integral de Neurociencias A.C., Móstoles, Madrid
  - Hospital 12 de Octubre, Madrid, Please Select
  - Hospital de La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid